CLINICAL TRIAL: NCT06871826
Title: Tissue Inhibitor of Metalloproteinases 2 Level Predicts Acute Kidney Injury in Patients Undergoing Cardiac Surgery
Brief Title: Tissue Inhibitor of Metalloproteinases 2 Level in Patients Undergoing Cardiac Surgery
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Wuhan University (Other)
Responsible Party: Principal Investigator, Jiahao Zhang, Department of Critical Care Medicine, Zhongnan Hospital of Wuhan University, Zhongnan Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 202123306
Record Dates: First submitted 2025-03-07; First posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Acute Kidney Injury; Extracorporeal Circulation; Complications; Surgery
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Intervention Model Description: TIMP2 level
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- TIMP2 Tertile 1 (Experimental): Other: TIMP2 level
  Interventions: Drug: TIMP2 level
- TIMP2 Tertile 2 (Experimental): Other: TIMP2 level
  Interventions: Drug: TIMP2 level
- TIMP2 Tertile 3 (Experimental): Other: TIMP2 level
  Interventions: Drug: TIMP2 level

INTERVENTIONS:
Drug: TIMP2 level — different TIMP2 level after on-pump cardiac surgery

SUMMARY:
Acute kidney injury (AKI) is one of the most frequent major complications in patients undergoing cardiac surgery. CSA-AKI is independently related to increased perioperative mortality, increased hospital and ICU length of stay as well as heath care expenditure. Identification of relevant biomarkers may lead to early diagnosis and improve patient outcomes and health care costs. The pathophysiology of CSA-AKI is complex and ischemia-reperfusion injury is one of the important factors. Recently, it has been shown that Tissue Inhibitor of Metalloproteinases 2 (TIMP2) is associated with ischemia-reperfusion injury. In this study, relationship between TIMP2 with the risk of CSA-AKI was analyzed and the predictive value of elevated level of TIMP2 for early prediction of CSA-AKI was further evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients (≥18 years old) underwent on-pump cardiac surgery
* admitted to ICU immediately after surgery

Exclusion Criteria:

* Patients younger than 18 years
* with prior AKI
* end-stage kidney disease
* need for chronic hemodialysis
* pregnant patients
* unable to give written consent for participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-07-22 (Actual); Primary Completion 2025-01-25 (Actual); Study Completion 2025-01-25 (Actual)

PRIMARY OUTCOMES:
the development of CSA-AKI | 1 Week
  the development of CSA-AKI

SECONDARY OUTCOMES:
AKI severity | 1 Week
  AKI stage 1，stage 2，stage 3
need for RRT | 1 Week
  Reflect kidney function
duration of AKI (≥7 days) | 1 Week
  Reflect kidney function
length of ICU stay | up to 28 days
  Reflect patient prognosis
post-operative hospital stay | up to 28 days
  Reflect patient prognosis

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongnan Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No